CLINICAL TRIAL: NCT02219815
Title: Pre-operative Rehabilitation for Reduction of Hospitalization After Coronary Bypass and Valvular Surgery.
Acronym: PREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Dr. Rakesh C. Arora, Medical Director, Intensive Care Cardiac Sciences, St. Boniface Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PREHAB
Record Dates: First submitted 2014-07-30; First posted 2014-08-19 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Patients Waiting for Coronary Artery Bypass Graft Surgery; Patients Waiting for Aortic Valve Repair or Replacement; Patients Waiting for Mitral Valve Repair or Replacement; Patients Waiting for Combined Procedures. (CAGB and Valve)
Keywords: Preoperative Care; Exercise Therapy; Cardiac Surgery; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): Patients in the standard care group will receive care as is currently delivered to patients awaiting cardiac surgery at each site. At present, patients are advised to rest and participate in very light intensity physical activity while awaiting surgery. At 1-2 weeks prior to their scheduled surgical date, the patient attends a single three hour cardiac pre-assessment with a nurse practitioner and cardiac anesthesiologist. In addition, a cardiac nurse counsels each patient on healthy behaviors (e.g. smoking cessation, diet, exercise).
- Prehab Intervention (Experimental): Patients in the Prehab group will receive, in addition to the standard of care, an eight-week comprehensive exercise therapy and education program at a community-based CR facility. Patients will be asked to complete at least two sessions of supervised, structured exercise class plus have the option to attend one additional exercise class per week for eight-weeks, with progression to a moderate to high-intensity interval program based on the supervised assessment of the patient's capabilities. Prehab participants will also attend four education sessions on topics such as risk factor reduction, medication use, cardiovascular physiology, smoking cessation, healthy eating, exercise, and stress management and promotion of self-managed care.
  Interventions: Behavioral: Prehab Intervention

INTERVENTIONS:
Behavioral: Prehab Intervention — Pre-operative, structured exercise intervention.
  Arms: Prehab Intervention

SUMMARY:
The PREHAB study is a clinical trial where frail patients waiting for heart surgery are randomly chosen to either receive the current standard of care or to participate in an 8-week exercise/education program at a community-based cardiac rehabilitation facility. Patients can wait for elective heart surgery for as long as 3-4 months. During this time, individuals are often fearful of making things worse, causing them to stop being active and further deteriorate their physical condition. This wait period presents a potential opportunity for health care providers to engage the patient to take control of their self-managed care prior to surgery with the intent of improving post-surgical outcomes. Patients randomized to the PREHAB intervention group will participate in supervised exercise twice per week in a program designed to improve physical functioning and exercise capacity. The investigators hypothesize that the PREHAB program for frail elderly patients awaiting an elective cardiac surgery will reduce frailty, improve exercise capacity, improve physical activity behaviour, improve in-hospital outcomes, improve clinical outcomes 3 months and 1 year postoperatively, and improve overall quality of life.

DETAILED DESCRIPTION:
PREHAB will be a three centre prospective, randomized, open, blinded endpoint (PROBE) controlled trial using assessor blinding and intention-to-treat analysis. The study will be conducted at three academic, tertiary care hospitals (St. Boniface Hospital, Winnipeg, MB, Montreal Heart Institute. Montreal QC and Queen Elizabeth II Health Sciences Centre, Halifax, NS) and one non-academic hospital (Saint John Regional Health Centre, Saint John, NB) that perform cardiac surgery. These sites were chosen based on similar patient populations and surgical waitlist times. Additionally, each of these sites are partnered with one or more community-based cardiac rehabilitation (CR) centres, which are certified medical fitness facilities dedicated to improving the health of the community through health promotion, disease prevention and rehabilitation services. These facilities offer expert guidance from certified professionals, innovative health enhancement programs, and provide integrated medical, rehabilitative and fitness services. The investigators intend to recruit a total of 244 participants to the study (122 per study arm), anticipating a 20% dropout rate to achieve an eventual sample size of 194 participants.

Patients in the PREHAB group will receive, in addition to standard of care, an eight-week comprehensive exercise therapy and education program at a community-based CR facility. This program will target both the physical and psycho-social-cognitive aspects of cardiac disease and frailty. In brief, participants will be required to complete an intake health status assessment by the CR team including a physiotherapist, cardiovascular nurse, and dietitian and complete a symptom-limited graded exercise stress test according to the American College of Sports Medicine Guidelines for Exercise Testing and Prescription 7th Edition. Patients will be asked to complete at least two sessions of supervised, structured exercise class plus have the option to attend one additional exercise class per week for eight-weeks, with progression to a moderate to high-intensity interval program based on the supervised assessment of the patient's capabilities. This has been shown to be safe and effective in unrepaired heart failure and elderly patients. PREHAB participants will also attend four education sessions on topics such as risk factor reduction, medication use, cardiovascular physiology, smoking cessation, healthy eating, exercise, and stress management and promotion of self-managed care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years and older, undergoing elective isolated coronary artery bypass grafting (CABG), aortic valve repair/replacement for moderate aortic stenosis or severe regurgitation, mitral valve repair/replacement for moderate stenosis or severe regurgitation or combined CABG/valve procedures
* Patients with Clinical Frailty Score (CFS) ≥3 (vulnerable) and < 7 (8 = very severely frail, approaching end-of-life or 9 = terminally ill) at time of acceptance for cardiac surgery
* Patients with an estimated ≥ 6 week wait time

Exclusion Criteria:

* Patients who have unstable or recent unstable cardiac syndrome as defined by:

  1. Severe heart failure (NYHA IV) or angina (CCS class IV) symptoms
  2. Critical left main (LM) coronary disease
  3. Hospitalization for arrhythmias, congestive heart failure or acute coronary syndrome prior to randomization
* Patients who have severe left ventricular obstructive disease as defined by:

  1. Severe aortic or mitral stenosis (aortic or mitral valve area <1.0cm2 or mean gradient > 40 mmHg or > 10 mmHg respectively)
  2. Dynamic left ventricular (LV) outflow obstruction
* Patients who have demonstrated exercise induced ventricular arrhythmias or have experienced a recent hospitalization for arrhythmias
* Patients who have cognitive deficits that would preclude rehabilitation
* Patients who have physical limitations that would preclude rehabilitation
* Patients who are unable to attend the Prehab program

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-04; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Arora, MD, Principal Investigator — St. Boniface Hospital/University of Manitoba
Locations (5):
- Canada (5):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Saint John Regional Hospital - New Brunswick Heart Centre, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Montreal Heart Institute, Montreal, Quebec
  - Laval University, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kehler DS, Stammers AN, Tangri N, Hiebert B, Fransoo R, Schultz ASH, Macdonald K, Giacomontonio N, Hassan A, Legare JF, Arora RC, Duhamel TA. Systematic review of preoperative physical activity and its impact on postcardiac surgical outcomes. BMJ Open. 2017 Aug 11;7(8):e015712. doi: 10.1136/bmjopen-2016-015712. PMID 28801404
- [Derived] Stammers AN, Kehler DS, Afilalo J, Avery LJ, Bagshaw SM, Grocott HP, Legare JF, Logsetty S, Metge C, Nguyen T, Rockwood K, Sareen J, Sawatzky JA, Tangri N, Giacomantonio N, Hassan A, Duhamel TA, Arora RC. Protocol for the PREHAB study-Pre-operative Rehabilitation for reduction of Hospitalization After coronary Bypass and valvular surgery: a randomised controlled trial. BMJ Open. 2015 Mar 9;5(3):e007250. doi: 10.1136/bmjopen-2014-007250. PMID 25753362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Prehab Intervention
Started | 44 | 45
Post Hospital Discharge Analysis (The study analysis for the primary outcome was based on this milestone. Post discharge is defined as completed surgery and discharged from hospital. This would complete the requirement for our analysis.) | 42 | 39
3 Month Post Surgery | 34 | 31
Completed | 22 | 21
Not Completed | 22 | 24

BASELINE CHARACTERISTICS:
Population: the baseline analysis was based on the completion of the primary outcome of hospital length of stay. Consented participants and participants in the analysis does differ. 8 participants were not involved in the analysis as they did not have surgery or had emergent surgery prior to intervention start.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Prehab Intervention | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 4 | 15
  >=65 years | 31 | 35 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (5.2) | 71.4 (6.4) | 70.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 31 | 34 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 42 | 39 | 81

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Hospital Length of Stay Greater Than 7 Days.
Description: Proportion of patients with hospital length of stay greater than 7 days compared to those with less than 7 days
Time Frame: Post-surgery (approximately 9 weeks after baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Prehab Intervention
Number analyzed (Participants) | 42 | 39
Participants | 20 | 16

2. Secondary Outcome: Baseline Exercise Capacity
Description: This measure will be assessed using the results of a 6 minute walk test.
Time Frame: baseline assessment - Study entry
Reporting Status: Not Posted

3. Secondary Outcome: Preoperative Exercise Capacity
Description: This measure will be assessed using the results of a 6 minute walk test.
Time Frame: Pre-Surgery (approximately 8 weeks after baseline)
Reporting Status: Not Posted

4. Secondary Outcome: 3-Month Exercise Capacity
Description: This measure will be assessed using the results of a 6 minute walk test.
Time Frame: 3 Months Post-Surgery (approximately 5 months after baseline)
Reporting Status: Not Posted

5. Secondary Outcome: 1-Year Exercise Capacity
Description: This measure will be assessed using the results of a 6 minute walk test.
Time Frame: 1 Year Post-Surgery (approximately 14 months after baseline)
Reporting Status: Not Posted

6. Secondary Outcome: Baseline Physical Activity Behaviour
Description: This measure will be assessed objectively using accelerometers. Moderate and vigorous physical activity (MVPA) will be compared
Time Frame: baseline assessment - Study entry
Reporting Status: Not Posted

7. Secondary Outcome: Preoperative Physical Activity Behaviour
Description: as for outcome 6
Time Frame: Pre-Surgery (approximately 8 weeks after baseline)
Reporting Status: Not Posted

8. Secondary Outcome: 3-Month Physical Activity Behaviour
Description: as for outcome 6
Time Frame: 3 Months Post-Surgery (approximately 5 months after baseline)
Reporting Status: Not Posted

9. Secondary Outcome: 1-Year Physical Activity Behaviour
Description: as for outcome 6
Time Frame: 1 Year Post-Surgery (approximately 14 months after baseline)
Reporting Status: Not Posted

10. Secondary Outcome: Baseline Health-Related Quality of Life
Description: This measure will be assessed using EuroQual-Visual Analogue Scale. (EQ-VAS) This scale ranges from 0 - 100 with 0 = worst health and 100 = best health
Time Frame: baseline assessment - Study entry
Reporting Status: Not Posted

11. Secondary Outcome: Preoperatve Health-Related Quality of Life
Description: as for outcome 10
Time Frame: Pre-Surgery (approximately 8 weeks after baseline)
Reporting Status: Not Posted

12. Secondary Outcome: 3-Month Health-Related Quality of Life
Description: as for outcome 10
Time Frame: 3 Months Post-Surgery (approximately 5 months after baseline)
Reporting Status: Not Posted

13. Secondary Outcome: 1-Year Health-Related Quality of Life
Description: as for outcome 10
Time Frame: 1 Year Post-Surgery (approximately 14 months after baseline)
Reporting Status: Not Posted

14. Secondary Outcome: Baseline Frailty
Description: This measure will be assessed using the Modified Fried Criteria score Score ranges from 0 - 5, 0=not frail, 1=prefrail, 2-5=frail
Time Frame: baseline assessment - Study entry
Reporting Status: Not Posted

15. Secondary Outcome: Preoperative Frailty
Description: as for outcome 14
Time Frame: Pre-Surgery (approximately 8 weeks after baseline)
Reporting Status: Not Posted

16. Secondary Outcome: 3-Month Frailty
Description: as for outcome 14
Time Frame: 3 Months Post-Surgery (approximately 5 months after baseline)
Reporting Status: Not Posted

17. Secondary Outcome: 1-Year Frailty
Description: This measure will be assessed using the Modified Fried Criteria Score ranges from 0 - 5, 0=not frail, 1=prefrail, 2-5=frail
Time Frame: 1 Year Post-Surgery (approximately 14 months after baseline)
Reporting Status: Not Posted

18. Secondary Outcome: Baseline Anxiety
Description: This measure will be assessed using the General Anxiety Disorder - 7 (GAD-7) Score is out of 0-21 points. The higher the score the more symptoms of anxiety may be observed
Time Frame: Baseline Assessment - Study entry
Reporting Status: Not Posted

19. Secondary Outcome: Preoperative Anxiety
Description: as for outcome 18
Time Frame: Pre-Surgery Assessment (approximately 8 weeks after baseline)
Reporting Status: Not Posted

20. Secondary Outcome: 3-Month Anxiety
Description: as for outcome 18
Time Frame: 3 Months Post-Surgery (approximately 5 months after baseline)
Reporting Status: Not Posted

21. Secondary Outcome: 1-Year Anxiety
Description: as for outcome 18
Time Frame: 1 Year Post-Surgery (approximately 14 months after baseline)
Reporting Status: Not Posted

22. Secondary Outcome: Baseline Depression
Description: This measure will be assessed using the Five-item Geriatric Depression Scale (GDS-5) Score is based from 0-5. A score of 2 or more may indicated symptoms of depression
Time Frame: Baseline Assessment - Study entry
Reporting Status: Not Posted

23. Secondary Outcome: Preoperative Depression
Description: as for outcome 22
Time Frame: Pre-surgery Assessment ( 8 weeks after baseline)
Reporting Status: Not Posted

24. Secondary Outcome: 3-Month Depression
Description: as for outcome 22
Time Frame: 3 Months Post-Surgery (approximately 5 months after baseline)
Reporting Status: Not Posted

25. Secondary Outcome: 1 Year Depression
Description: as for outcome 22
Time Frame: 1 year Post-Surgery (approximately 14 months after baseline)
Reporting Status: Not Posted

26. Secondary Outcome: Postoperative Major Adverse Events
Description: Major adverse events include death, myocardial infarction (MI), stroke or renal failure requiring dialysis.
Time Frame: Post-Surgery (approximately 9 weeks after baseline)
Reporting Status: Not Posted

27. Secondary Outcome: Postoperative Cardiac Rehabilitation Attendance
Description: Will be assessed using administrative data from participating cardiac rehabilitation facilities.
Time Frame: Post-Surgery (approximately 20 weeks after baseline)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard Care | Prehab Intervention
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/42 | 1/39
Other Adverse Events (participants affected / at risk) | 8/42 | 3/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=42) | Prehab Intervention (N=39)
Stroke (Vascular disorders) | 2 (2) | 1 (1) — Patient suffered a stroke post surgery
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=42) | Prehab Intervention (N=39)
post operative Delirium (Nervous system disorders) | 8 (8) | 3 (3)

LIMITATIONS AND CAVEATS:
1. Recruitment was only 89 participants from an expected sample size of 244 participants. This was a major limitation regarding data analysis.
2. Short cardiac surgery waitlists (i.e. surgery in less than 4 weeks) were impactful to study recruitment and intervention delivery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT02219815/Prot_SAP_000.pdf
  • Informed Consent Form (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT02219815/ICF_001.pdf